CLINICAL TRIAL: NCT05579782
Title: Assessing Benefits of NIRAF Detection for Identifying Parathyroid Glands During Total Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Vanderbilt University (Other)
Responsible Party: Principal Investigator, Tracy S. Wang, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00040573
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Hypoparathyroidism; Thyroid Disease; Thyroid Neoplasms; Thyroid Cancer
MeSH Terms: conditions — Thyroid Diseases; Thyroid Neoplasms

STUDY DESIGN:
Intervention Model Description: NIRAF detection technology is used as an adjunctive tool for intraoperative parathyroid identification in patients who undergo total thyroidectomy (TTx) with or without lymph node dissection (LND) in the interventional group.
  Generic Name of Device: Parathyroid Autofluorescence Detection Device (NIRAF detection technology).
  The Parathyroid Autofluorescence Detection Device consists of a disposable fiber-optic probe that emits non-ionizing radiation from a NIR 785 nanometer (nm) laser source, and also transmits the resulting tissue NIRAF to a photo detector. The 785 nm laser source emits a maximum power of 20 Milliwatts (mW). The device has an FDA clearance for clinical use in general surgeries and dermatological use (Class 2 device).
Who Masked: Participant
Masking Description: Only participants will be masked to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- NIRAF Detection Technology (+) (Experimental): Parathyroid gland identification will be performed with PTeye using NIRAF detection technology as an adjunctive tool in patients who undergo total thyroidectomy (TTx) with or without lymph node dissection (LND).
  Interventions: Device: NIRAF Detection Technology
- NIRAF Detection Technology (-) (No Intervention): Parathyroid gland identification will be performed by the surgeon using only visual identification and without using PTeye - NIRAF detection technology in patients who undergo total thyroidectomy (TTx) with or without lymph node dissection (LND).

INTERVENTIONS:
Device: NIRAF Detection Technology — Near Infrared Autofluorescence (NIRAF) detection technology or 'PTeye' consists of a disposable fiber-optic probe that emits non-ionizing radiation from a NIR 785 nm laser source, and also transmits the resulting tissue NIRAF to a photo detector. The 785 nm laser source emits a maximum power of 20 mW. The device is FDA cleared for clinical use in general surgeries and dermatological use (Class 2 device).
  After surgeon identifies a potential parathyroid gland in the surgical field, the surgeon places the fiber-optic probe of PTeye on suspect tissue and presses the device foot-pedal to activate tissue NIRAF measurement. Auditory beep at high frequency with a Detection Ratio > 1.2 is interpreted by device as the suspect tissue being positive for parathyroid.
  Other Name: PTeye Device
  Arms: NIRAF Detection Technology (+)

SUMMARY:
This study describes a single center, randomized, single-blinded clinical trial to assess the clinical benefits of the use of near infrared autofluorescence (NIRAF) detection with an FDA-cleared device 'Parathyroid Eye (PTeye)' for identifying parathyroid glands during total thyroidectomy. It compares risk-benefits and outcomes in patients undergoing total thyroidectomy where NIRAF detection with PTeye for parathyroid identification is either used or not used.

DETAILED DESCRIPTION:
Inadvertent damage or excision of a healthy parathyroid gland (PG) following a total thyroidectomy (TTx) could result in transient hypocalcemia (< 6 months) in 5 - 35% of cases or permanent hypocalcemia (> 6 months) in 7% of the patients (1, 2). In both of these circumstances, patients would require calcium and active vitamin D supplementation in addition to a potentially prolonged hospital stay and/or unplanned hospital readmission adding to unnecessary burden and healthcare costs. These complications could be minimized with label-free intraoperative PG identification using near infrared autofluorescence (NIRAF) detection with a fiber-probe based approach as utilized in 'PTeye', which is medical device that was recently FDA-cleared. However, the true impact of this particular NIRAF-based approach on patient outcomes is yet to be determined

The aim of this prospective single blinded randomized study is to compare 2 groups of patients: TTx patients operated using NIRAF detection technology with PTeye as adjunct tool (NIRAF+) vs. patients operated without the adjunct technology (NIRAF-). The main objective of this study is to assess the benefit of intraoperative use of NIRAF detection technology via PTeye during TTx procedures with regard to postoperative hypocalcemia, PG identification, PG auto-transplantation and inadvertent resection rates compared to standard of care.

ELIGIBILITY:
Inclusion Criteria:

(i) All patients eligible for total thyroidectomy (TTx), with or without lymph node dissection. (includes patients undergoing a TTx who have undergone a prior neck exploration for parathyroid disease or other but have an intact thyroid).

(ii) All patients undergoing completion thyroidectomy.

Exclusion Criteria:

(i) Patients with concurrent parathyroid disease.

(ii) Patients with incidental enlarged parathyroid discovered during TTx.

(iii) Patients undergoing thyroid lobectomy/partial thyroidectomy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy S Wang, MD, MPH, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cousart AG, Kiernan CM, Willmon PA, Thomas G, Wang TS, Gauger PG, Duh QY, Underwood HJ, Jackson A, Patel A, Mahadevan-Jansen A, Solorzano CC. Near-Infrared Autofluorescence for Parathyroid Detection During Endocrine Neck Surgery: A Randomized Clinical Trial. JAMA Surg. 2025 Sep 1;160(9):936-944. doi: 10.1001/jamasurg.2025.2233. PMID 40668552

RESULTS

PARTICIPANT FLOW:
Groups:
- NIRAF Detection Technology (+): Parathyroid gland identification will be performed with PTeye using NIRAF detection technology as an adjunctive tool in patients who undergo total thyroidectomy (TTx) with or without lymph node dissection (LND).
  NIRAF Detection Technology: Near Infrared Autofluorescence (NIRAF) detection technology or 'PTeye' consists of a disposable fiber-optic probe that emits non-ionizing radiation from a NIR 785 nm laser source, and also transmits the resulting tissue NIRAF to a photo detector. The 785 nm laser source emits a maximum power of 20 mW. The device is FDA cleared for clinical use in general surgeries and dermatological use (Class 2 device).
  After surgeon identifies a potential parathyroid gland in the surgical field, the surgeon places the fiber-optic probe of PTeye on suspect tissue and presses the device foot-pedal to activate tissue NIRAF measurement. Auditory beep at high frequency with a Detection Ratio > 1.2 is interpreted by device as the suspect tissue being positive for parathyroid.
  Other Name: PTeye Device
Period: Overall Study
Arm/Group | NIRAF Detection Technology (+) | NIRAF Detection Technology (-)
Started | 39 | 41
Completed | 39 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NIRAF Detection Technology (+) | NIRAF Detection Technology (-) | Total
Number analyzed (Participants) | 39 | 41 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 30 | 61
  >=65 years | 8 | 11 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 29 | 56
  Male | 12 | 12 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 32 | 32 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 39 | 41 | 80

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Transient Hypoparathyroidism.
Description: The number of subjects with hypoparathyroidism. For the transient hypoparathyroidism; the definition utilized was a serum parathyroid hormone (PTH) level <10 pg/mL.
Time Frame: 24-48 hours post-op
Measure: Count of Participants; unit: Participants
Arm/Group | NIRAF Detection Technology (+) | NIRAF Detection Technology (-)
Number analyzed (Participants) | 39 | 41
Participants | 10 | 14

2. Primary Outcome: Patients With Hypoparathyroidism at Last Follow-up
Description: The number of subjects with hypoparathyroidism at last follow-up. Follow-up defined as PTH less than the normal institutional range.
Time Frame: 2 days to 1 year after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | NIRAF Detection Technology (+) | NIRAF Detection Technology (-)
Number analyzed (Participants) | 39 | 41
Participants | 1 | 1

3. Secondary Outcome: Overall Average Number of Parathyroid Glands Identified With High Confidence.
Description: Overall number of parathyroid glands identified (Experimental Group: Glands identified with naked eye + NIRAF; Control Group: Glands identified with naked eye)
Time Frame: Immediate (during total thyroidectomy, up to 3 hours)
Measure: Mean (95% Confidence Interval); unit: Number of parathyroid glands
Arm/Group | NIRAF Detection Technology (+) | NIRAF Detection Technology (-)
Number analyzed (Participants) | 39 | 41
Number of parathyroid glands | 3.4 [3.2 to 3.7] | 2.9 [2.5 to 3.2]

4. Secondary Outcome: Number of Participants With Frozen Sections Sent for Analysis.
Description: Number of participants with frozen sections sent for analysis during the procedure to confirm potential parathyroid tissue.
Time Frame: Immediate (during total thyroidectomy, up to 3 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | NIRAF Detection Technology (+) | NIRAF Detection Technology (-)
Number analyzed (Participants) | 39 | 41
Participants
  0 frozen sections | 38 | 30
  greater than or equal to 1 frozen sections | 1 | 11

5. Secondary Outcome: Number of Participants With Auto-transplanted Parathyroid Glands
Description: Number of participants with auto-transplanted parathyroid glands if the parathyroid gland was accidentally excised/devascularized.
Time Frame: Immediate (during total thyroidectomy, up to 3 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | NIRAF Detection Technology (+) | NIRAF Detection Technology (-)
Number analyzed (Participants) | 39 | 41
Participants
  o auto-transplanted parathyroid glands | 31 | 31
  1 auto-transplanted parathyroid glands | 7 | 8
  greater than or equal to 2 auto-transplanted parathyroid glands | 1 | 2

6. Secondary Outcome: Number of Participants Who Spent Nights in the Hospital After Total Thyroidectomy
Description: Number of participants who spent nights for postoperative recovery in the hospital after the surgical procedure.
Time Frame: 0-72 hours after total thyroidectomy
Measure: Count of Participants; unit: Participants
Arm/Group | NIRAF Detection Technology (+) | NIRAF Detection Technology (-)
Number analyzed (Participants) | 39 | 41
Participants
  0 nights | 0 | 1
  1 night | 39 | 38
  more than one night | 0 | 2

7. Secondary Outcome: Number of Participants With Inadvertently Resected Parathyroid Glands
Description: Number of participants with inadvertently resected parathyroid glands when parathyroid tissue is found in the resected thyroid specimens.
Time Frame: Immediate (intraoperative) to 7-10 days after total thyroidectomy (pathology report)
Measure: Count of Participants; unit: Participants
Arm/Group | NIRAF Detection Technology (+) | NIRAF Detection Technology (-)
Number analyzed (Participants) | 39 | 41
Participants | 9 | 8

8. Secondary Outcome: Number of Doctor Visits/Emergency Department Visits or Hospital Admissions
Description: Number of doctor visits/emergency department visits or hospital admissions due to hypocalcemia and or associated symptoms.
Time Frame: Up to 6 months after total thyroidectomy
Measure: Number; unit: Number of events
Arm/Group | NIRAF Detection Technology (+) | NIRAF Detection Technology (-)
Number analyzed (Participants) | 39 | 41
Number of events | 0 | 0

9. Secondary Outcome: Duration and Total Daily Dosage of Calcium and/or Vitamin D Supplementation After Surgery
Description: Duration and total daily dosage of calcium and/or vitamin D supplementation after surgery - if patient had no prior history of supplementation.
Time Frame: Up to 6 months after total thyroidectomy
Population: We would not be able to provide precise data regarding duration and total daily dosage. Following surgery, those at risk for hypocalcemia are prescribed calcium standing dose and patients are also counseled to take additional calcium supplements. It is not possible to calculate an exact dose. Patients often take calcium supplements. Therefore, the additional calcium and the exact duration of when they stopped additional calcium is challenging for patients and was not collected in the trial.
Arm/Group | NIRAF Detection Technology (+) | NIRAF Detection Technology (-)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | NIRAF Detection Technology (+) | NIRAF Detection Technology (-)
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/41
Other Adverse Events (participants affected / at risk) | 0/39 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-31): https://cdn.clinicaltrials.gov/large-docs/82/NCT05579782/Prot_SAP_002.pdf
  • Informed Consent Form (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT05579782/ICF_001.pdf